CLINICAL TRIAL: NCT06788574
Title: Preliminary Outcome Of Tecar Therapy Effect On Stress Urinary Incontinence, Pelvic Floor Strength And Sexual Satisfaction In Women Complaining Of Vaginal Relaxation Syndrome: A Randomized Controlled Trial
Brief Title: Preliminary Outcome Of Tecar On Stress Urinary Incontinence, Pelvic Floor Strength And Sexual Satisfaction In Women With Vaginal Relaxation Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Magdy Ahmed, Department of Physical therapy for Women Health, Faculty of Physical therapy, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (P.T.WH/3/2021/9).
Record Dates: First submitted 2025-01-08; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: STRESS URINARY INCONTINENCE; VAGINAL RELAXATION SYNDROME
Keywords: Vaginal Relaxation Syndrome; Tecar Therapy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tecar group (Experimental): consists of 20 females who will receive TECAR therapy and PFM exercises
  Interventions: Device: TECAR device: MCRR. The sign producer is an INDIBA® 448 kHz RF device that has a vaginal/ or rectum electrode (made in Barcelona, Spain); Procedure: pelvic floor exercises
- Control group (Sham Comparator): consist of 20 females who will receive sham tecar and PFM exercises
  Interventions: Procedure: pelvic floor exercises; Device: Sham device

INTERVENTIONS:
Device: TECAR device: MCRR. The sign producer is an INDIBA® 448 kHz RF device that has a vaginal/ or rectum electrode (made in Barcelona, Spain) — TECAR (Transfer Electrical, Capacitive, and Resistive) is originally used in Italy. TECAR therapy is a radiofrequency (RF) therapy, which produces high-frequency waves. RF can be capacitive or resistive The capacitive mode (CET) generates energy in electrolyte-rich soft tissues such as muscles and vascular or lymphatic tissues . The resistive mode (RET) directs energy to deeper tissues that contain more fat and fibers (such as bones, ligaments, and tendons;
  Arms: Tecar group
Procedure: pelvic floor exercises — pelvic floor exercise will be performed with the perineometer twice a week for eight weeks (16 sessions), with five sets of 20 repetitions each
Device: Sham device — sham treatment by Tecar device for 15 min without producing any waves.
  Arms: Control group

SUMMARY:
Forty women aged 50-60 years with a body mass index (BMI) of 25 kg/m2 to 30 kg/m2, who complain of stress urinary incontinence and vaginal laxity, will be separated randomly into two equivalent groups. In group (A) 20 women will receive TECAR therapy for 15 min and pelvic floor exercise for 20 min, while in group (B), 20 females will receive sham treatment for 15 min and pelvic floor exercise for 20 min twice per week for 8 weeks. Both groups wil be assessed using a perineometer as an assessment tool for pelvic floor muscle strength muscles and the Visual Analog Scale, ICIQ-UI short form questionnaire about the frequency of urinary incontinence symptoms, Millheiser Sexual Satisfaction Scale, and the Sexual Quality of Life Questionnaire-Female (SQOL-F) to assess sexual satisfaction by each patient before, after 4 weeks, and after 8 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* participants are multipara at least two times with sexual activity for at least 1/month with normal cell cytology (PAP smear), integrity of the vaginal canal mucosa, and negative urine culture (without injuries or bleeding).

Exclusion Criteria:

* pregnancy, use of photosensitive medicines, vaginal bleeding injury or infection in the treated area, and use of an IUD.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women who complain of stress urinary incontinence and vaginal laxity
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
pelvic floor muscle strength assessed using a Peritron (9300) device with a vaginal sensor | after 4 and 8 weeks
  At baseline and after 4 and 8 weeks for each female in both groups will be assessed using a Peritron (9300) device with a vaginal sensor (Peritron 9300). Cardio Design Pty, Australia designed Peritron 9300. Description in technical terms: 0-300 cm H2o numerical data, 1 cm H2o resolution, 1 cm H2o accuracy for 95% of data, 3.5 digits liquid crystal panel, 12.7 mm high with a battery charge indication vaginal probe, 28 mm in diameter, and 30 mm in length
urinary incontinence symptoms using Visual Analog Scale and ICIQ-UI short form questionnaire | after 4 and 8 weeks
  using Visual Analog Scale and ICIQ-UI short form questionnaire The visual analogue scale (VAS) is a rating tool will be used to graphically evaluate the severity of a patient's reported urinary incontinence symptoms. The patient will instructed to cross the VAS by uniformly spacing numerical values along a 10-centimeter line.
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence
sexual satisfaction using Millheiser Sexual Satisfaction Scale, and the Sexual Quality of Life Questionnaire-Female (SQOL-F) | after 4 and 8 weeks
  Millheiser Sexual Satisfaction Scale, and the Sexual Quality of Life Questionnaire-Female (SQOL-F) Millheiser sexual satisfaction scale 1 = None, 2 = Poor, 3 = Fair, 4 = Good, 5 = Very good, 6 = Excellent (Millheiser et al., 2010).
  The Sexual Quality of Life-Female (SQOL-F) questionnaire is a short instrument that specifically assesses the relationship between female sexual dysfunction and quality of life. It consists of 18 items, rated using a six-point scale (completely agree to completely disagree).Each item on the scale is scored between 1 and 6 (1 = I completely agree, 2 = I mostly agree, 3= I partially agree, 4 = I partially do not agree, 5= I mostly disagree, 6 = I completely disagree).
Vaginal PH using PH color strips | at baseline, after 4 weeks, and after 8 weeks of treatment
  PH color strips will be used to assess vaginal PH for each woman in both groups (A and B) at baseline, after 4 weeks, and after 8 weeks of treatment (orange = 5, yellow = 6, light green = 7, dark green= 8, blue petroleum = 9; Kulp et al., 2008).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://doi.org/10.3389/fpsyg.2022.1062363